CLINICAL TRIAL: NCT02995993
Title: An Open-Label, Multi-Center Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Moss-aGal in Patients With Fabry Disease
Brief Title: Pharmacokinetics, Pharmacodynamics, and Safety of Moss-aGalactosidase A in Patients With Fabry Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Greenovation Biotech GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CT-GR-MaGal-01
Record Dates: First submitted 2016-12-14; First posted 2016-12-19 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moss-aGal (Experimental): Single administration of 0.2 mg/kg recombinant human alpha-galactosidase A produced in moss (moss-aGal) as intravenous infusion
  Interventions: Drug: Moss-aGal (recombinant human alpha-galactosidase A produced in moss)

INTERVENTIONS:
Drug: Moss-aGal (recombinant human alpha-galactosidase A produced in moss) — Single i.v. Infusion of 0.2 mg/kg moss-aGal over 60 minutes

SUMMARY:
Six patients with Fabry disease will be recruited. Patients will receive a single dose of 0.2 mg/kg recombinant human alpha-galactosidase A produced in moss (moss-aGal) as intravenous infusion. Patients will be hospitalized during the infusion and for at least 24 hours after the end of the infusion. Treatment will be administered sequentially: if a patient shows no safety concerns on the treatment day, treatment of the next patient will commence on the following day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Fabry disease evidenced by a deficient α-galactosidase A (α-Gal A) activity or an α-Gal A gene mutation (the latter is mandatory in women);
* Treatment naïve Fabry patients or Fabry patients who paused any enzyme replacement therapy for Fabry disease due to personal reasons for 3 months before study entry;
* Female and male patients between 18 and <=65 years;
* At least one of the clinical manifestations of Fabry disease including neuropathic pain, angiokeratoma, cornea verticillata, cardiomyopathy, hypo- or anhydrosis, abdominal pain, diarrhea, serum creatinine >1.0 mg/dL, or proteinuria >300 mg/24 hours;
* Lyso-Gb3 concentrations in plasma above upper limit of normal;
* Male patients with a female partner of child-bearing potential agree to use a medically acceptable method of contraception (e.g. condoms, sexual abstinence, vasectomy), not including the rhythm method for 30 days after administration of the study medication;
* Female patients of childbearing potential must apply a highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly [e.g. implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, or a vasectomized partner]). The birth control method must have been applied for at least one monthly cycle prior to the first administration of study medication and 30 days after administration of the study medication.
* Patient is willing and able (in the opinion of the investigator) to understand and comply with the procedures and evaluations of the study;
* Patient must be willing and legally able to give written informed consent.

Exclusion Criteria:

* Treatment with any enzyme replacement therapy for Fabry disease within 3 months before study entry;
* Fabry patients who paused any enzyme replacement therapy for Fabry disease due to intolerability;
* Patient is positive for anti-alpha-Gal A immunoglobulin G (IgG) at Screening;
* Participation in any other clinical study with a medical device or investigational medicinal product concurrently or within 3 months before study start;
* Patient is currently on dialysis, is expected to begin dialysis during the study, has received a kidney transplant, or is on the renal transplant waiting list;
* Patient is unable to comply with the protocol (e.g. clinical relevant medical condition making implementation of the protocol difficult, unstable social situation, or otherwise unlikely to complete the study) or is, in the opinion of the investigator, otherwise unsuited for the study;
* Known human immunodeficiency virus, hepatitis B surface antigen and/or hepatitis C infection;
* Known allergies or intolerabilities to enzyme replacement therapy;
* Hypersensitivity (like anaphylactic reaction) to the active substance or to any excipients of moss-aGal;
* Co-administration of moss-aGal with chloroquine, amiodarone, benoquin or gentamicin;
* Breast-feeding and pregnant women;
* Patients with liver impairment;
* Women with signs of cardiac fibrosis detectable by echocardiography;
* Other, not Fabry disease-related severe illnesses;
* Malignancies within the past 5 years;
* Liver transaminases >=3 times above the upper Limit of normal;
* Alcohol and/or drug abuse;
* Weight >100 kg;
* Employees of the sponsor or patients who are employees or relatives of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | PK sampling for 24 h after moss-aGal administration
  Area under the serum concentration curve extrapolated to infinity
Number of patients with drug-related adverse events | Adverse event monitoring for 28 days after moss-aGal administration

SECONDARY OUTCOMES:
Gb3 concentration in plasma | Monitoring up to Day 28 after moss-aGal administration
  Globotriaosylceramide concentration in plasma
Gb3 concentration in morning urine | Monitoring up to Day 28 after moss-aGal administration
  Globotriaosylceramide concentration in morning urine
Lyso-Gb3 concentration in plasma | Monitoring up to Day 28 after moss-aGal administration
  Globotriaosylsphingosine concentration in plasma

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Ruhruniversität Bochum, Klinik für Kinder- und Jugendmedizin im St. Josef-Hospital im Katholischen Klinikum Bochum, Bochum
  - Universitätsmedizin Mainz, Zentrum für Kinder- und Jugendmedizin, Mainz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen JS, Busch A, Day TS, Meng XL, Yu CI, Dabrowska-Schlepp P, Fode B, Niederkruger H, Forni S, Chen S, Schiffmann R, Frischmuth T, Schaaf A. Mannose receptor-mediated delivery of moss-made alpha-galactosidase A efficiently corrects enzyme deficiency in Fabry mice. J Inherit Metab Dis. 2016 Mar;39(2):293-303. doi: 10.1007/s10545-015-9886-9. Epub 2015 Aug 27. PMID 26310963